CLINICAL TRIAL: NCT03822429
Title: Cumulative Live Birth Rate (CLBR) After a Complete IVF Cycle: a Single Center
Brief Title: Cumulative Live Birth Rate (CLBR) After a Complete IVF Cycle: a Single Center Retrospective Study
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: ART; Fertility Disorders
Keywords: CLBR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- women < 35 years old
  Interventions: Drug: Controlled ovarian stimulation
- women between 36 and 38 years old
  Interventions: Drug: Controlled ovarian stimulation
- women between 39 and 40 years
  Interventions: Drug: Controlled ovarian stimulation
- women > 41 years old
  Interventions: Drug: Controlled ovarian stimulation

INTERVENTIONS:
Drug: Controlled ovarian stimulation — Hormonal therapy to induce ovulation by multiple ovarian follicles

SUMMARY:
We need to identify a new parameter to evaluate the success rate of IVF techniques. CLBR has been suggested as a suitable way for reporting success of IVF program: it implies capturing the totality of live birth episodes following successive treatments. For patients CLBR is easy to understand because it summarizes the chance of a live birth over an entire treatment period. CLBR per oocyte retrieval is more meaningful as it is the best indicator of quality and success in IVF and it allows the best indicator of quality and success in IVF with different strategies for freezing embryos.

DETAILED DESCRIPTION:
Traditionally, studies about In Vitro Fertilization (IVF) examine and report the 'per cycle' and 'per embryo transfer procedure' probability of pregnancy and delivery .Thus, each IVF cycle is considered as a unique entity even if several embryo transfers (ET) have been performed after a single ovarian stimulation.

Thanks to the latest technological refinements, in recent years the number of thawed frozen ETs has greatly increased and has become an essential feature of IVF procedures .This practice has been encouraged by the strategy of preferring single ET for reducing multiple pregnancy and preventing ovarian hyperstimulation in high risk women.

Moreover, at first infertility counseling patients usually want to know which is their possibility to have a live birth child with ART treatment, after the first stimulation cycle, also involving the chances after frozen ET or frozen oocytes injection.

Live birth rate (LBR) after a single fresh or frozen ET appears, at present time, to be an insufficient parameter for a realistic evaluation of the efficacy of an IVF program.

We need to identify a new parameter for the evaluation of the success rate of IVF techniques which should incorporate outcomes associated with a single controlled ovarian stimulation cycle. Specifically, Cumulative live birth rate (CLBR) has been suggested as a suitable way for reporting success of IVF program : it implies capturing the totality of live birth episodes following successive treatments.

For patients CLBR is very reliable and easy to understand because it summarizes the chance of a live birth over an entire treatment period . CLBR per oocyte retrieval is more meaningful as it is the best indicator of quality and success in IVF and it allows the best indicator of quality and success in IVF with different strategies for freezing embryos.

The aim of the present study was to report our experience on CLBR after the first stimulation cycle and to determinate which prognostic factors contribute to positive pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Humanitas Research hospital for undergoing their first IVF cycle

Exclusion Criteria:

* cycle with any pre-implatation genetic test

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients admitted to Humanitas Research hospital for undergoing their first IVF cycle , except cycle with any pre-implatation genetic test
Sampling Method: Non-Probability Sample
Enrollment: 6375 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative Live Birth Rate | 2 years
  number of live Birth derived from a complete controlled ovarian stimulation

IPD SHARING:
Plan to Share IPD: No